CLINICAL TRIAL: NCT03553420
Title: Osse Registry for Patients With Lipodystrophy Run by the European Consortium of Lipodystrophies (ECLip)
Brief Title: Registry for Patients With Lipodystrophy
Acronym: ECLip Registry
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Collaborators: Sorbonne University (Other); University Hospital, Lille (Other); University of Cambridge (Other); Endocrinology Research Centre, Moscow (Other Government); University of Leipzig (Other); University of Amsterdam (Other); Dokuz Eylul University (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); University of Rome Tor Vergata (Other); University of Pisa (Other); University of Santiago de Compostela (Other); Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other); University Hospital Muenster (Other); Szeged University (Other); Centro Hospitalar do Porto (Other); University Medical Centre Ljubljana (Other); Medical University of Vienna (Other); National and Kapodistrian University of Athens (Other); Stoffwechselzentrum St. Gallen (Unknown); National Taiwan University Hospital (Other); Marmara University (Other); University of Palermo (Other); Attikon Hospital (Other); Kinderkrankenhaus auf der Bult (Other); Hopital Universitaire Robert-Debre (Other); University of Milan (Other); C.I. Parhon National Institute of Endocrinology (Other)
Responsible Party: Principal Investigator, Julia von Schnurbein, Prinicipal Investigator, University of Ulm
Other Study IDs: ECLip Registry
Record Dates: First submitted 2018-03-14; First posted 2018-06-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Lipodystrophy Acquired; Lipodystrophy Congenital
Keywords: lipodystrophy
MeSH Terms: conditions — Lipodystrophy, Familial Partial; Lipodystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Given the lack of knowledge on lipodystrophies, the medical and social responsibility for the persons affected by it calls for the monitoring of the progression over long periods of time. Sensible clinical and basic research into rare diseases such as lipodystrophy is only possible in multi-location networks with sufficient case numbers. Also, reliable information on the incidence of certain manifestation patterns, health status, etc. is of utmost importance for health care and health policy in this rare disease.

Therefore, the European Consortium of Lipodystrophies (ECLip), an association of European experts on lipodystrophy, has launched a registry (OSSE) for lipodystrophies which is committed to help to improve the research conditions by consolidating this kind of information in a registry.

DETAILED DESCRIPTION:
As lipodystrophies are rare diseases subdivided into yet rarer sub-groups, research in this field requires international co-operation.

The European Consortium of Lipodystrophy (ECLip) consists of an association of European experts in the field of lipodystrophy. It has set up a Registry Board to implement a registry for patients with lipodystrophy using the Open Source Software OSSE (Open Source Registry System for Rare Diseases in the EU), which is a web based platform focused on a federated approach that allows to perform distributed searches which are designed to comply data protection requirements and preserve data sovereignty. To ensure data protection, medical and identifying data will be stored on two different servers both run by the Institute for Epidemiology and Medical Biometry of the University of Ulm.

Medical centers from all over the world where patients are treated with lipodystrophy are invited to join the ECLip Registry and to become ECLip Registry members. Upon registration, they can enter patient data after they have obtained local ethic committee permission and the patient in question has given written consent to this. Data entry is done at the individual locations via a web-based user interface. Identifying data are recorded directly into the identity management system. Communication between the identity management and the OSSE registry happens via a web browser.

The aim of the patient registry is to compile data on the natural history of each different sub-group of lipodystrophies, their comorbidities, treatment options used and medical and quality of life out-come for the patients. For this, the following data retrieved from regular patient visits are collected:

* Precise diagnosis including moleculargenetic results
* Clinical presentation and comorbidities
* Laboratory changes and results of diagnostic procedures
* Natural course of the disease including age at onset of disease and comorbidities
* Family history

Research within this registry can be performed by participating clinicians/researchers and third parties after a research proposal has be accepted by the responsible committee of the ECLip. The registry aims to answer the following questions

* new insights into the pathophysiology of lipodystrophy
* improve therapeutic options for the patients
* compile information material for patients, families and relevant professionals

ELIGIBILITY:
Inclusion Criteria:

* lipodystrophy

Exclusion Criteria:

* lipodystrophy due to anti-retroviral drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with lipodystrophy not due to anti-retroviral drugs presenting to a participating center might be entered
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-12-16 (Actual); Primary Completion 2068-01 (Estimated); Study Completion 2068-01 (Estimated)

PRIMARY OUTCOMES:
Age at death | after 20 years
  patients are followed regularly, age at death (years) will be documented

SECONDARY OUTCOMES:
change in somatic comorbidities under standard treatment | yearly for 50 years
  standardized physical examination, laboratory and instrument based tests
genotype-phenotype correlation for patients with familial lipodystrophy | every 5 years for 50 years
  molecular genetic results will be compared to results from standardized physical examination, laboratory and instrument based tests
age at onset of metabolic complications | yearly for 50 years
  metabolic complications will be assessed via standardized physical examination, laboratory and instrument based tests
age at onset orthopedic complications | yearly for 50 years
  orthopedic complications will be assessed via standardized physical examination, laboratory and instrument based tests
age at onset neuromuscular complications | yearly for 50 years
  neuromuscular complications will be assessed via standardized physical examination, laboratory and instrument based tests

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wabitsch, Prof. Dr., Study Chair — University of Ulm; David Araujo-Vilar, Prof. Dr., Principal Investigator — Santiago de Compostela University; Julia von Schnurbein, Dr., Principal Investigator — University of Ulm; Gabriele Nagel, Prof., Principal Investigator — University of Ulm; Camille Vatier, Dr., Principal Investigator — Pierre et Marie Curie School of Medicine (Paris); Marie-Christine Vantyghem, Prof., Principal Investigator — Lille University; Giovanni Ceccarini, Dr., Principal Investigator — Endocrine Unit, University Hospital of Pisa; David Savage, Prof., Principal Investigator — University of Cambridge Metabolic Research Laboratories
Locations (28):
- Medical University of Vienna, Vienna, Austria
- France (3):
  - Lille University, Lille
  - AP-HP Nord Université de Paris, Hôpital Universitaire Robert-Debré, Paris
  - Pierre et Marie Curie School of Medicine, Sorbonne University, Paris
- Germany (4):
  - Kinder-und Jugendkrankenhaus AUF DER BULT, Hanover
  - Department of Internal Medicine (Endocrinology and Nephrology), University of Leipzig, Leipzig
  - Med. Klinik B für Gastroenterologie und Hepatologie, Universitätsklinikum Münster, Münster
  - Dept for Pediatrics and Adolescent Medicine, University of Ulm: Interdisciplinary obesity clinic, Ulm
- Greece (2):
  - National and Kapodistrian University of Athens, Athens
  - Second Department of Internal Medicine, Medical School, National and Kapodistrian University of Athens, Attikon University Hospital, Athens
- University of Szeged, Department of Internal Medicine, Szeged, Hungary
- Italy (6):
  - Endocrinology Unit, Department of Clinical and Medical science, S. Orsola-Malpighi Hospital , University of Bologna, Bologna
  - Policlinic University Hospital of Milan, Milan
  - Universita del piemonte Orientale, Novara
  - Palermo University, Palermo
  - Endocrine Unit of University Hospital of Pisa, Pisa
  - Tor Vergata University - Policlinico of Tor Vergata, Roma
- Academic Medical Center, University of Amsterdam, Amsterdam, Netherlands
- Abel Salazar Biomedical Sciences Institute - University of Porto, Porto, Portugal
- C. I. Parhon National Institute of Endocrinology, Bucharest, Romania, Bucharest, Romania
- Endocrinology Research Centre, Moscow, Russia
- University Medical Center Ljubljana - Clinical Institute of Medical Genetics, Ljubljana, Slovenia
- Santiago de Compostela University, Santiago de Compostela, Spain
- Stoffwechselzentrum friendlydocs, Sankt Gallen, Switzerland
- National Taiwan University Hospital, Taipei, Taiwan
- Turkey (Türkiye) (2):
  - Marmara University, Pediatric Endocrinology and Diabetes, Istanbul
  - Dokuz Eylul University School of Medicine, Izmir
- University of Cambridge Metabolic Research Laboratories, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researches participating in the ECLip registry and third parties independently can request to perform research with the data.
Time Frame: As soon as data is entered into the registry, request for data analysis can be handed in.
Access Criteria: Researchers participating in the ECLip registry and independent third parties can request to perform research with the data. For this a formal request for data analysis (data evaluation form; available from the Registry Board) has to be handed to the leader of the Registry Board who will pass it to all board members. These will form a proposal for the Registry members.
URL: https://www.eclip-web.org/information/registry/

REFERENCES:
- [Background] von Schnurbein J, Adams C, Akinci B, Ceccarini G, D'Apice MR, Gambineri A, Hennekam RCM, Jeru I, Lattanzi G, Miehle K, Nagel G, Novelli G, Santini F, Santos Silva E, Savage DB, Sbraccia P, Schaaf J, Sorkina E, Tanteles G, Vantyghem MC, Vatier C, Vigouroux C, Vorona E, Araujo-Vilar D, Wabitsch M. European lipodystrophy registry: background and structure. Orphanet J Rare Dis. 2020 Jan 15;15(1):17. doi: 10.1186/s13023-020-1295-y. PMID 31941540